CLINICAL TRIAL: NCT01711476
Title: Influence of Meal Timing on Glucose Metabolism and Hyperandrogenism in Lean Women With Polycystic Ovary Syndrome
Brief Title: Meal Timing on Glucose and Hyperandrogenism in PCOS Women
Acronym: MealTimePCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas Caracas (Other)
Responsible Party: Principal Investigator, Daniela Jakubowicz, MD, MD, Hospital de Clinicas Caracas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCCCBI 018-2008-104
Record Dates: First submitted 2012-10-17; First posted 2012-10-22 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Polycystic Ovary Syndrome (PCOS) Women
Keywords: PCOS; Bdiet; Ddiet; OGTT
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling ARM 1 (Active Comparator): Arm 1 Breakfast Diet The arm 1 will be assigned to eat High calorie breakfast (800kcal) and reduced dinner (200 kcal) During 90 days from baseline to the end of the trial (day 90)
  Interventions: Other: Active Comparator: Lifestyle counseling ARM 1
- Lifestyle counseling ARM 2 (Placebo Comparator): Lean PCOS women in the Arm 2 will be assigned to do a dinner diet from day 0 to day 90 of the trial
  Interventions: Behavioral: Placebo Comparator: Lifestyle counseling Dinner Diet ARM 2

INTERVENTIONS:
Behavioral: Placebo Comparator: Lifestyle counseling Dinner Diet ARM 2 — In this Arm 2 group the PCOS will be assigned to dinner diet and we will compare the androgen levels Day 0 to androgen after DAY 90 of this diet also we will compare Glucose and Insulin response to OGTT Day 0 and Day 90, and ovulatory frequency along alll the 90 days of the Dinner diet
  Other Names: The lean PCOS patients assigned to dinner diet
  Arms: Lifestyle counseling ARM 2
Other: Active Comparator: Lifestyle counseling ARM 1 — In the Arm 1 we will measure androgen levels and insulin and glucose response to OGTT at baseline DAY 0 and after 90 days on the dinner diet (Day 90) for comparison Also we will evaluate by weekly progesterone the ovulatory events
  Other Names: Lean PCOS women in ARM 1 will be assigned to Breakfast diet from Day 0 to day 90 of the study
  Arms: Lifestyle counseling ARM 1

SUMMARY:
The objective of this study is to investigate the effects of two isocaloric maintenance diets with different meal timing distribution on insulin resistance hyperandrogenism and cytochrome P450c17 alpha activity in lean PCOS women.

The investigators hypothesis is that in lean PCOS women a Breakfast Diet (BD) which consist in high calorie breakfast and reduced dinner, vs Dinner Diet (DD) which consist in high calorie dinner with reduced breakfast; the BD will improve glucose and insulin response to OGTT and would decrease the hyperandrogenism and cytochrome P450c17 alpha activity.

DETAILED DESCRIPTION:
Hyperinsulinemia plays a central role in the pathogenesis in obese as well as in lean PCOS women. These women are insulin resistant and have compensatory hyperinsulinemia that stimulates ovarian cytochrome P450c17 alpha activity that in turn stimulates ovarian androgen concentrations.

In obese PCOS women, weight loss improves insulin resistance and hyperandrogenism, resulting in improvement of clinical symptoms.

Since lean PCOS women do not have the option of weight loss, it is important to know if composition and meal timing distribution may influence glucose metabolism and hyperandrogenism and cytochrome P450c17 alpha activity. We hypothesized that a timing pattern of increased nutrient intake of protein and carbohydrates in the morning, with decreased caloric intake at night would improve insulin sensitivity and hyperandrogenism in lean women with PCOS

ELIGIBILITY:
Inclusion Criteria:

lean women with Polycystic Ovary BMI below 25 kg/m2 Testosterone above 1.0 ng/ml 17 Oh progesterone below 200 ng/ml US of Polycystic Ovaries

Exclusion Criteria:

Obesity BMI above 25 kg/m2 Diabetes Mellitus Other endocrine disease like hypothyroidism, late onset adrenal hyperplasia Pregnancy Contraceptive or other hormonal treatment

Ages: 22 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Androgens and 17 alpha hydroxyprogesterone serum levels | 90 days
  The androgens (testosterone, free testosterone, DHEA-S, androstenedione)and 17 alpha hydroxyprogesterone will be measured at baseline and again will be measured at the end of the trial by day 90. In both groups or Arms one on breakfast diet and the other on dinner diet.

SECONDARY OUTCOMES:
Glucose and Insulin Response to OGTT | 90
  Glucose and Insulin Response to OGTT will be measured at baseline and again will be repeated after 90 days of the trial for comparison One group will be assigned to breakfast diet and the other group to dinner diet

OTHER OUTCOMES:
Ovulatory frequency | 90 days
  From baseline (day O) to the end of the study (day 90) progesterone will be quantified weekly to assess the ovulation in both of the group (The ovulation in the breakfast diet group will be compared to that of the dinner diet group)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Jakubowicz, MD, Principal Investigator — Hospital de Clinicas Caracas
Locations (1):
- Daniela Jakubowicz, Caracas, San Bernardino, Venezuela